CLINICAL TRIAL: NCT02841410
Title: Neural Networks of Decision Making Processes Triggered by Food Labels
Brief Title: Neuroeconomic Approach of Food Nutritionnal Assesment
Acronym: NeuroFood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC14.322
Record Dates: First submitted 2016-07-05; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteer
Keywords: Food; Emotion; Health; Nutrition; Heuristic; Reasoning; Magnetic Resonance Imaging
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteer (Other)
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging

SUMMARY:
This fMRI study evaluated the cognitive mechanisms and the cerebral substrate of decision making when evaluating the healthiness of food products with nutritional information displayed either with a Traffic Light system, a colored nutritional label, and a Guideline Daily Amount system, a numeric label.

DETAILED DESCRIPTION:
The investigators postulated that Traffic Light label would recruit emotion processes and activation of subjacent cerebral networks.

On the contrary, the nutritional information presented in a Guideline Daily Amount label, would recruit, due to its numeric format and higher complexity, supplementary cognitive processes and activation of related brain regions.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* medical exam completed before participation in reserach
* to be insured under the social security system
* to be an adult between 18 and 50 years

Exclusion Criteria:

* counter-argument to magnetic field exposure
* neurological or psychiatric disorder including eating disorders
* had

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of cerebral areas's activation | About two hours
  MRI

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Krainik, Principal Investigator — Grenoble Hospital University

REFERENCES:
- [Background] Arana FS, Parkinson JA, Hinton E, Holland AJ, Owen AM, Roberts AC. Dissociable contributions of the human amygdala and orbitofrontal cortex to incentive motivation and goal selection. J Neurosci. 2003 Oct 22;23(29):9632-8. doi: 10.1523/JNEUROSCI.23-29-09632.2003. PMID 14573543
- [Background] Aschemann-Witzel J, Grunert KG, van Trijp HC, Bialkova S, Raats MM, Hodgkins C, Wasowicz-Kirylo G, Koenigstorfer J. Effects of nutrition label format and product assortment on the healthfulness of food choice. Appetite. 2013 Dec;71:63-74. doi: 10.1016/j.appet.2013.07.004. Epub 2013 Jul 23. PMID 23891558
- [Background] Basten U, Biele G, Heekeren HR, Fiebach CJ. How the brain integrates costs and benefits during decision making. Proc Natl Acad Sci U S A. 2010 Dec 14;107(50):21767-72. doi: 10.1073/pnas.0908104107. Epub 2010 Nov 30. PMID 21118983
- [Background] Beaver JD, Lawrence AD, van Ditzhuijzen J, Davis MH, Woods A, Calder AJ. Individual differences in reward drive predict neural responses to images of food. J Neurosci. 2006 May 10;26(19):5160-6. doi: 10.1523/JNEUROSCI.0350-06.2006. PMID 16687507
- [Background] Birch LL. Development of food preferences. Annu Rev Nutr. 1999;19:41-62. doi: 10.1146/annurev.nutr.19.1.41. PMID 10448516
- [Background] Borgmeier I, Westenhoefer J. Impact of different food label formats on healthiness evaluation and food choice of consumers: a randomized-controlled study. BMC Public Health. 2009 Jun 12;9:184. doi: 10.1186/1471-2458-9-184. PMID 19523212
- [Background] Braeutigam S, Rose SP, Swithenby SJ, Ambler T. The distributed neuronal systems supporting choice-making in real-life situations: differences between men and women when choosing groceries detected using magnetoencephalography. Eur J Neurosci. 2004 Jul;20(1):293-302. doi: 10.1111/j.1460-9568.2004.03467.x. PMID 15245501
- [Background] Burton S, Andrews JC. (1996), Age, Product Nutrition, and Label Format Effects on Consumer Perceptions and Product Evaluations. Journal of Consumer Affairs, 30, 68-89.
- [Background] Campos S, Doxey J, Hammond D. Nutrition labels on pre-packaged foods: a systematic review. Public Health Nutr. 2011 Aug;14(8):1496-506. doi: 10.1017/S1368980010003290. Epub 2011 Jan 18. PMID 21241532
- [Background] Carelli RM, King VC, Hampson RE, Deadwyler SA. Firing patterns of nucleus accumbens neurons during cocaine self-administration in rats. Brain Res. 1993 Oct 29;626(1-2):14-22. doi: 10.1016/0006-8993(93)90557-4. PMID 8281424
- [Background] De Neys W, Glumicic T. Conflict monitoring in dual process theories of thinking. Cognition. 2008 Mar;106(3):1248-99. doi: 10.1016/j.cognition.2007.06.002. Epub 2007 Jul 12. PMID 17631876
- [Background] De Neys W, Vartanian O, Goel V. Smarter than we think: when our brains detect that we are biased. Psychol Sci. 2008 May;19(5):483-9. doi: 10.1111/j.1467-9280.2008.02113.x. PMID 18466410
- [Background] Frackowiak RSJ, Friston KJ, Frith C, Dolan R, Price CJ, Zeki S, Ashburner J, Penny WD. (2003). Human Brain Function. Academic Press, 2nd edition
- [Background] Frank S, Kullmann S, Veit R. Food related processes in the insular cortex. Front Hum Neurosci. 2013 Aug 23;7:499. doi: 10.3389/fnhum.2013.00499. eCollection 2013. PMID 23986683
- [Background] Friston KJ, Ashburner J, Kiebel SJ, Nichols TE, Penny WD. (2007). Statistical Parametric Mapping: The Analysis of Functional Brain Images. Academic Press
- [Background] Goel V. Anatomy of deductive reasoning. Trends Cogn Sci. 2007 Oct;11(10):435-41. doi: 10.1016/j.tics.2007.09.003. Epub 2007 Oct 2. PMID 17913567
- [Background] Goel V, Dolan RJ. Explaining modulation of reasoning by belief. Cognition. 2003 Feb;87(1):B11-22. doi: 10.1016/s0010-0277(02)00185-3. PMID 12499108
- [Background] Grabenhorst F, Schulte FP, Maderwald S, Brand M. Food labels promote healthy choices by a decision bias in the amygdala. Neuroimage. 2013 Jul 1;74:152-63. doi: 10.1016/j.neuroimage.2013.02.012. Epub 2013 Feb 18. PMID 23428568
- [Background] Grimm O, Jacob MJ, Kroemer NB, Krebs L, Vollstadt-Klein S, Kobiella A, Wolfensteller U, Smolka MN. The personality trait self-directedness predicts the amygdala's reaction to appetizing cues in fMRI. Appetite. 2012 Jun;58(3):1023-9. doi: 10.1016/j.appet.2012.02.007. Epub 2012 Feb 28. PMID 22381514
- [Background] Grunert KG, Wills JM, Fernandez-Celemin L. Nutrition knowledge, and use and understanding of nutrition information on food labels among consumers in the UK. Appetite. 2010 Oct;55(2):177-89. doi: 10.1016/j.appet.2010.05.045. Epub 2010 May 28. PMID 20546813
- [Background] Hare TA, Camerer CF, Rangel A. Self-control in decision-making involves modulation of the vmPFC valuation system. Science. 2009 May 1;324(5927):646-8. doi: 10.1126/science.1168450. PMID 19407204
- [Background] Hsu M, Bhatt M, Adolphs R, Tranel D, Camerer CF. Neural systems responding to degrees of uncertainty in human decision-making. Science. 2005 Dec 9;310(5754):1680-3. doi: 10.1126/science.1115327. PMID 16339445
- [Background] Kahneman D, Tversky A. (1973). On the psychology of prediction. Psychological Review, 80, 237-251.
- [Background] Kahneman, D., Tversky, A. (1979). Prospect theory: An analysis of decisions under risk. Econometrica, 47, 263-291.
- [Background] Knutson B, Rick S, Wimmer GE, Prelec D, Loewenstein G. Neural predictors of purchases. Neuron. 2007 Jan 4;53(1):147-56. doi: 10.1016/j.neuron.2006.11.010. PMID 17196537
- [Background] Loewenstein GF, Weber EU, Hsee CK, Welch N. Risk as feelings. Psychol Bull. 2001 Mar;127(2):267-86. doi: 10.1037/0033-2909.127.2.267. PMID 11316014
- [Background] Loewenstein GF, Lerner JS. (2003). The role of affect in decision making. In Handbook of Affective Sciences. RJ Davidson, KR Scherer, HH Goldsmith, eds. Oxford: Oxford University Press, 619-42.
- [Background] McClure SM, Li J, Tomlin D, Cypert KS, Montague LM, Montague PR. Neural correlates of behavioral preference for culturally familiar drinks. Neuron. 2004 Oct 14;44(2):379-87. doi: 10.1016/j.neuron.2004.09.019. PMID 15473974
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Background] Rozin P, Ashmore M, Markwith M. Lay American conceptions of nutrition: dose insensitivity, categorical thinking, contagion, and the monotonic mind. Health Psychol. 1996 Nov;15(6):438-47. doi: 10.1037//0278-6133.15.6.438. PMID 8973924
- [Background] Siep N, Roefs A, Roebroeck A, Havermans R, Bonte ML, Jansen A. Hunger is the best spice: an fMRI study of the effects of attention, hunger and calorie content on food reward processing in the amygdala and orbitofrontal cortex. Behav Brain Res. 2009 Mar 2;198(1):149-58. doi: 10.1016/j.bbr.2008.10.035. Epub 2008 Nov 6. PMID 19028527
- [Background] Simon, D., Holyoak, K.J. (2002). Structural dynamics of cognition: From consistency theories to constraint satisfaction. Personality and Social Psychology Review, 6, 283-294.
- [Background] Slovic, P., Finucane, M., Peters, E., MacGregor, D.G. (2002). The affect heuristic. In: Gilovich, T., Griffin, D., Kahneman, D. (Eds.), Heuristics and Biases: The Psychology of Intuitive Judgment. Cambridge University Press, New York, pp. 397-420.
- [Background] Tiger, L. (1992). The pursuit of pleasure. Boston, MA: Little, Brown
- [Background] Tsujii T, Watanabe S. Neural correlates of belief-bias reasoning under time pressure: a near-infrared spectroscopy study. Neuroimage. 2010 Apr 15;50(3):1320-6. doi: 10.1016/j.neuroimage.2010.01.026. Epub 2010 Jan 18. PMID 20080190
- [Background] von Neumann, J., Morgenstern, O. (1944). Theory of Games and Economic Behavior, Princeton University Press.
- [Background] Yokum S, Ng J, Stice E. Attentional bias to food images associated with elevated weight and future weight gain: an fMRI study. Obesity (Silver Spring). 2011 Sep;19(9):1775-83. doi: 10.1038/oby.2011.168. Epub 2011 Jun 16. PMID 21681221
- [Background] Zajonc, R.B. (1980). Feeling and thinking: Preferences need no inferences. American Psychologist, 35, 151-175.